CLINICAL TRIAL: NCT02251834
Title: Hispanic Secondary Stroke Prevention Initiative
Acronym: HISSPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Olveen Carrasquillo, Olveen Carrasquillo, MD, MPH, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20140423; R01MD009164 (NIH)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: Healthcare Disparities; stroke; Hispanic Americans; community health worker; Mobile Health; Transient Ischemic Attack (TIA); hypertension; Randomized Controlled Trial; high cholesterol; behavioral; exercise; diabetes; diet
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Hypertension; Hypercholesterolemia; Behavior; Motor Activity; Diabetes Mellitus | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Health Worker (Experimental): Community Health Worker (CHW) home visits, coaching phone calls, group sessions .
  Interventions: Behavioral: Community Health Worker (CHW)
- Usual Care (Other): usual care and health education brochures every 4 months.
  Interventions: Other: usual care and health education brochures every 4 months.

INTERVENTIONS:
Behavioral: Community Health Worker (CHW) — The primary mechanism used by the Community Health Worker (CHW) for delivering interventions will be a) home visits b) phone based contacts c) group level activities d) mobile technology. Ideally, each subject will have, at a minimum, 4 home visits and ten phone calls during months 3-12. Group visits will held twice a month. The Community Health Worker (CHW) intervention will be highly individualized and tailored to unique circumstances of each patient and we expect home visits, calls, ProMobile usage and group visits to vary by patient.
  Arms: Community Health Worker
Other: usual care and health education brochures every 4 months. — Patients randomized to the control group will receive usual care.
  Arms: Usual Care

SUMMARY:
Stroke is a leading cause of death and functional impairments and stroke risk factors (SRFs) disproportionately affect Latino populations. In the Hispanic Secondary Stroke Prevention Initiative (HISSPI) the investigators propose a study using Community Health Workers (CHW) and mobile technologies using cell phones to reduce the risk for a recurrent stroke among Latino stroke patients.

The project examines the effectiveness of a combined multilevel intervention consisting of Community Health Workers (CHW) and mobile based phone technologies in lowering of systolic blood pressure (SBP) which is the most important risk factor for recurrent stroke.

DETAILED DESCRIPTION:
Stroke is the fourth leading cause of death, and the main cause of adult disability in the US. As the population ages, over the next 3 decades the number of strokes is expected to double. At the same time, the Hispanic population, currently the largest minority group in the US is expected to double. The rapid growth and aging of Hispanics will lead to dramatic future increases in the public health impact of stroke. This group of investigators and others have extensively described the disproportionate burden of stroke and stroke risk factors (SRFs) (e.g. blood pressure, diabetes, and lipids) among Hispanics. Over the last two decades, community health workers (CHWs) have emerged as one of the more promising strategies at addressing Latino health disparities. However, evidence from randomized controlled trials (RCTs) supporting this approach remains limited. Recent technology based interventions, particularly those using mobile-based platforms (e.g. phone text messaging), have shown tremendous potential at improving outcomes among minority populations. This team's ongoing line of investigation is testing Community Health Workers (CHWs) interventions through rigorous randomized controlled trials (RCTs) aimed at improving clinical outcomes for a variety of health conditions including diabetes, cancer and Human Immunodeficiency Virus (HIV) disease. The investigators are also leading several studies addressing ProMobile technologies among minority elders. To date, preliminary data suggests each of these two approaches independently may lead to considerable improvements in some stroke risk factors (SRFs). However, evidence for the use of these combined approaches from studies using rigorous experimental designs for most health conditions has been limited. Further, data on these promising interventions among Hispanic stroke patients remains a major gap in the field of stroke disparities.

In the Hispanic Secondary Stroke Prevention Intervention (HISSPI),the investigators propose a translational research study addressing minority health in the form of a pragmatic clinical trial aimed at improving health outcomes among Latinos. The project extends their ongoing work with Community Health Workers (CHWs) and mobile phone technologies to examine the effectiveness of this combined multilevel intervention as an adjunct to routine health care targeting stroke risk factors (SRFs) among Hispanic patients having had a recent stroke. The investigators focus on this group of patients because they have an over 25% risk of recurrent stroke in the next five years, with the second stroke often being much more debilitating than the first stroke.

The study will be conducted at two hospitals in Miami-Dade county (one public, one private). With a highly diverse Latino population, both Caribbean and Central/South Americans, Miami is an ideal laboratory to test such an approach in an immigrant community facing numerous distinct barriers to quality stroke care. Hispanic Secondary Stroke Prevention Initiative (HISPPI) also leverages existing resources, including those of the recently funded Florida Puerto Rico Collaboration to Reduce Stroke Disparities and the Clinical Translational Science Award (CTSA). The investigators expect this translational research to provide new insights on approaches that can transform medical practice and improve health outcomes in Latino populations; particularly, in the context of ongoing reforms in health care delivery. The study design is a randomized controlled trial (RCT) of 300 Latino stroke patients admitted with an ischemic or hemorrhagic stroke, having a minimal to moderate disability as a result of the stroke but whom are ambulatory modified Rankin Scale (mRS) <=3.

Primary Objectives: Based on evidence based guidelines to prevent a recurrent stroke, the investigators will determine if the proposed intervention results in improved systolic blood pressure among the intervention versus usual care group. Blood pressure management is the single most important risk factor for preventing a recurrent stroke.

Secondary Objectives: The investigators will also examine if the proposed intervention results in improvements in other secondary stroke risk factors including low density lipoprotein, adherence to statin therapy,adherence to antiplatelet/anti-thrombotic therapy, and among patients with diabetes, better glycemic control.

Additional outcomes: As hypothesis generating analyses, the investigators will examine, the following outcomes:

1. Quality of Life
2. Health Care utilization (visits to primary care providers and stroke specialists)
3. Proportion of patients re-hospitalized for recurrent stroke

Hypotheses: Consistent with guidelines on systolic blood pressure (SBP) reductions that would lead to clinically meaningful reductions in recurrent stroke risk, the investigators hypothesize that at 12 months, as compared to usual care, patients randomized to the Community Health Worker (CHW) ProMobile intervention will have a systolic blood pressure that is 8mmHg lower. Least detectable differences for secondary outcomes: With 300 patients, the investigators will have over 80% power to detect differences in intervention versus control group of 1) Low-density lipoprotein (LDL) that is 13ml/dl lower 2) 15% greater adherence to statin and antiplatelet/thrombotic therapy 3) among the subset having diabetes, glycated haemoglobin (HbA1c) that is 0.9% lower.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* History of an ischemic or intra-cerebral hemorrhagic stroke within the past five years
* Be Hispanic/Latino on self report
* modified Rankin Scale (mRs) ≤ 3
* Reside in Miami-Dade County

Exclusion Criteria:

* Any life-threatening morbidity including an active cancer diagnosis
* Enrollment in other non acute stroke, cardiovascular, diabetes study
* Patients with an arm circumference of ≥47 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | one year
  Our primary hypothesis is that at twelve months, patients in the intervention arm will have SBP on average, 8mmHg lower than those in the control group.

SECONDARY OUTCOMES:
LDL | one year
  Achieving an LDL-C level of 70 mg/dL is associated with a 28% stroke risk reduction and stroke patients with a 50% reduction in LDL-C had a 35% reduction in combined risk of nonfatal and fatal stroke.
Self-reported adherence to statins and anti-platelet medications | one year
  Morisky medication adherence scale
A1C | one year
  among patients having diabetes we will measure A1C

CONTACTS AND LOCATIONS:
Overall Officials: Olveen Carrasquillo, MD, MPH, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Carrasquillo O, Young B, Dang S, Fontan O, Ferras N, Romano JG, Dong C, Kenya S. Hispanic Secondary Stroke Prevention Initiative Design: Study Protocol and Rationale for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Oct 19;7(10):e11083. doi: 10.2196/11083. PMID 30341050